CLINICAL TRIAL: NCT03368833
Title: Caudal Blockade and Electrocardiographic Changes
Status: Terminated | Type: Observational
Why Stopped: Caudal blockade no longer being used in the ORs at this hospital.
Sponsor: Senthil G. Krishna (Other)
Responsible Party: Sponsor-Investigator, Senthil G. Krishna, Attending Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB17-00861
Record Dates: First submitted 2017-09-28; First posted 2017-12-11 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Regional Anesthesia Morbidity
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caudal block: Patients that receive regional anesthesia in the form of a caudal block prior to surgery as part of their standard of care.
  Interventions: Diagnostic Test: Electrocardiogram
- Control: Patients who do not receive a caudal block.
  Interventions: Diagnostic Test: Electrocardiogram

INTERVENTIONS:
Diagnostic Test: Electrocardiogram — 12-lead ECG will be obtained after induction and at 5, 10, 20, 30, and 60 minutes after the caudal epidural block.
  Other Names: ECG; EKG

SUMMARY:
Caudal epidural blockade is frequently used as an adjunct to general anesthesia in children for perioperative analgesia. Intravascular injection of local anesthetic is a known complication that can adversely affect the neurological and cardiovascular systems. This study will look at the delayed effects of a caudal epidural block on the electrical activity of the patient's myocardium by trying to characterize the incidence of ECG changes within 60 minutes after the caudal dose is given.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade 1 or 2
* Receiving general anesthesia with a caudal block

Exclusion Criteria:

* Preexisting cardiac comorbidities

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients having general surgery at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Change in T wave amplitude | Baseline to 60 mins. post caudal
  Change in T wave amplitude on the ECG tracings
Change in T wave width | Baseline to 60 mins. post caudal
  Change in T wave width on the ECG tracings

CONTACTS AND LOCATIONS:
Overall Officials: Senthil Krishna, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No